CLINICAL TRIAL: NCT06579742
Title: A Clinical Trial to Examine the Efficacy of a Supplement to Support Healthy Hair and Skin
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scale Media Inc (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20423
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Hair Thinning; Hair Loss
Keywords: Skin Aging; Loss of Skin Elasticity; Skin Health; Hair Health
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live Conscious Beyond Collagen Supplement (Experimental): Participants in this arm will receive the Live Conscious Beyond Collagen supplement. The supplement contains Vitamin C (90 mg), Biotin (2500 mcg), and a Proprietary Collagen Blend (10.1 g) including Types I & III Bovine Collagen, Type II Marine Collagen, Type II Chicken Sternum Collagen, and Types I, V & X Eggshell Membrane Collagen.
  Interventions: Dietary Supplement: Live Conscious Beyond Collagen
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo product. The placebo contains Maltodextrin.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Live Conscious Beyond Collagen — Participants in the experimental arm will take 1 scoop (10.4 g) of Live Conscious Beyond Collagen supplement mixed with 12 fl oz of water in the evening after their last meal of the day for 24 weeks.
  Arms: Live Conscious Beyond Collagen Supplement
Dietary Supplement: Placebo — Participants in the placebo comparator arm will take 1 scoop (10.4 g) of the placebo product (Maltodextrin) mixed with 12 fl oz of water in the evening after their last meal of the day for 24 weeks.
  Arms: Placebo

SUMMARY:
This is a triple-blinded, randomized, placebo-controlled clinical trial designed to evaluate the efficacy of Scale Media's Live Conscious Beyond Collagen supplement on overall hair and skin health. The study will involve 50 male or female participants aged 40 and over who have self-perceived hair thinning and shedding. The trial will last for 24 weeks and includes the completion of questionnaires and photo submissions at specific time points.

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* Self-perceived hair thinning, specifically on the top and crown of the scalp for at least three months
* Self-perceived increased hair shedding for at least three months
* Concerns regarding skin health and appearance
* Has been using the same hair care routine and products for at least one month prior to the study, i.e., shampoo, conditioner, and products
* Has been using the same skincare routine and products for at least one month prior to the study, i.e., moisturizer, serums, etc.
* Willing to maintain the same hair care routine and products throughout the study
* Willing to maintain the same skincare routine and products throughout the study
* Willing to maintain the same diet and exercise regimen during the study
* Willing to refrain from taking any vitamins, minerals, or herbal supplements that target hair growth or skin health during the study
* Willing to refrain from taking any new vitamins, minerals, or supplements of any kind during the study
* Willing to avoid introducing any new prescription medications or supplements that target hair health and appearance of skin health and appearance during the study
* Be generally healthy and do not live with any uncontrolled chronic disease
* Willing to stop taking any other multivitamin supplements at least one month prior to and for the entire study duration
* Willing to avoid dyeing the hair for the duration of the study
* Living with someone who can take their study photos for the duration of the study

Exclusion Criteria:

* Anyone with a diagnosed hair loss or hair thinning health condition, except for female pattern baldness (e.g., alopecia areata)
* Women who are pregnant, breastfeeding, or trying to conceive
* Anyone currently taking iron supplements
* Anyone unwilling or unable to follow the study protocol
* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
* Anyone who does not consume animal products for personal or religious reasons
* Is undergoing or planning to undergo laboratory testing and/or significant medical procedures during the study duration
* A history of severe allergic reactions, including but not limited to any of the product's ingredients
* Has undergone any chemical treatments to the hair in the last three months, e.g., chemical straightening, hair extensions with chemical bonding, perms, and relaxers
* Has any planned chemical treatments for the hair during the study period, e.g., chemical straightening, hair extensions with chemical bonding, perms, and relaxers
* Has any planned cosmetic treatments to the face, including botox, dermal filler, chemical peels, etc.
* Currently undergoing hair loss treatment, including mechanical scalp stimulation, or has done so in the last three months
* Currently using other hair growth/thickening products
* Currently taking any prescription medication for hair loss, or has done so in the last three months
* Currently taking any prescription medication for skin health, or has done so in the last three months
* Has undergone any surgeries or invasive treatments in the last six months
* Has had any major illness in the last three months
* Currently taking medication that has hair loss as a known or observed side effect
* Currently undergoing or have you recently undergone chemotherapy or radiotherapy
* Anyone who has had a hair transplant within the last year

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hair Density and Hair Volume | Baseline, Month 3, and Month 6
  Hair health will be assessed through expert dermatologist grading and participant questionnaires to measure changes in hair density and hair volume over the course of the study.

SECONDARY OUTCOMES:
Change in Skin Health (Fine Lines, Wrinkles, Texture, and Elasticity) | Baseline, Month 3, and Month 6
  Skin health will be evaluated using participant self-reported questionnaires and expert dermatologist grading to assess changes in fine lines, wrinkles, skin texture, elasticity, brightness, radiance, firmness, and roughness over the course of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No